CLINICAL TRIAL: NCT02073383
Title: Prospective Randomized Study of Three Different Techniques for Ultrasound Guided Axillary Brachial Plexus Block
Brief Title: Three Techniques for Ultrasound Guided Axillary Brachial Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FUSaoPaulo - USG Guided Block
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Hand Surgery
Keywords: Axillary brachial plexus block; Ultrasound; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Around Artery (Experimental): Intervention Name: Axillary brachial plexus block
  Group A: 30 ml of 0.375% bupivacaine will be injected around the artery . If this were a clock, would deposit 7,5 ml of anesthetic in positions 0, 3, 6 and 9 .
  Interventions: Procedure: Axillary brachial plexus block
- Two injections (Experimental): Group 2: 30 ml of bupivacaine 0.375 % below the artery will be injected in the 6 o'clock position .
  Interventions: Procedure: Axillary brachial plexus block
- Perineural (Active Comparator): Group Perineural : 10 ml of bupivacaine 0.375 % will be injected around the median, ulnar and radial nerves .
  Interventions: Procedure: Axillary brachial plexus block

INTERVENTIONS:
Procedure: Axillary brachial plexus block

SUMMARY:
The brachial plexus block is an anesthetic technique often used for surgical procedures of the upper limb. The brachial plexus block through the axilla (BPVA) is one of the techniques most commonly used to obtain regional anesthesia of the upper limbs, being performed by anesthesia of the terminal branches of the brachial plexus, which would be the ulnar, median, radial and musculocutaneous nerves. With the aid of ultrasound , two techniques can be used to perform the BPVA . The first , known as multiple puncture technique , the local anesthetic is deposited around each nerve that want to block . This technique is most commonly used to perform the BPVA . The second technique , known as 2 injections , local anesthetic is deposited below the axillary artery and around the musculocutaneous nerve . This technique has been proposed to try to reduce the execution time of anesthesia . Studies actually show that the technique of 2 injections showed less time to perform the block, with the same success rate. However, the technique of 2 injections showed a longer latency and higher rate of vascular puncture . (14) In order to perform a procedure with shorter execution time , without changing the latency, success rate and ensuring patient safety , the investigators designed this protocol to evaluate three techniques for performing the ultrasound- guided axillary brachial plexus block.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the patient (IC)
* Indication for brachial plexus block for anesthesia and analgesia in candidates for hand surgical procedures
* ASA physical status I, II or III according to the American Association of Anesthesiology.

Exclusion Criteria:

* Cognitive impairment or psychiatric disease
* Active infection condition at the puncture site of the block
* Bleeding disorders
* History of allergy to bupivacaine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-12 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to compare the efficacy of the three different techniques for ultrasound guided axillary brachial plexus block | The primary outcome will be measured at the same day of the procedure.
  The brachial plexus block is performed through the axilla , with the aid of ultrasound and a peripheral nerve stimulator with the patient in the supine position. The needle that will be used is 22G x 50 mm . After disinfection and skin antisepsis with chlorhexidine , tha puncture site will be infiltrated with 1% lidocaine . Furthermore, musculocutaneous nerve will be blockade with 10 ml of 0.375% bupivacaine for all patients. Patients will be divided into three groups :
  Group A: 30 ml of 0.375% bupivacaine will be injected around the artery . If this were a clock, would deposit 7,5 ml of anesthetic in positions 0, 3, 6 and 9 .
  Group 2 injections : 30 ml of bupivacaine 0.375 % below the artery will be injected in the 6 o'clock position .
  Group M : 10 ml of bupivacaine 0.375 % will be injected

SECONDARY OUTCOMES:
Block Latency | 30 minutes
  Latency time of the blockade , defined as the time between the end of injection of local anesthetic will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Thompson GE, Rorie DK. Functional anatomy of the brachial plexus sheaths. Anesthesiology. 1983 Aug;59(2):117-22. doi: 10.1097/00000542-198308000-00009. PMID 6869868
- [Background] Klaastad O, Smedby O, Thompson GE, Tillung T, Hol PK, Rotnes JS, Brodal P, Breivik H, Hetland KR, Fosse ET. Distribution of local anesthetic in axillary brachial plexus block: a clinical and magnetic resonance imaging study. Anesthesiology. 2002 Jun;96(6):1315-24. doi: 10.1097/00000542-200206000-00009. PMID 12170042
- [Background] DE JONG RH. Axillary block of the brachial plexus. Anesthesiology. 1961 Mar-Apr;22:215-25. doi: 10.1097/00000542-196103000-00010. No abstract available. PMID 13720553
- [Background] Vester-Andersen T, Christiansen C, Sorensen M, Kaalund-Jorgensen HO, Saugbjerg P, Schultz-Moller K. Perivascular axillary block II: influence of injected volume of local anaesthetic on neural blockade. Acta Anaesthesiol Scand. 1983 Apr;27(2):95-8. doi: 10.1111/j.1399-6576.1983.tb01913.x. PMID 6837255
- [Background] Groban L. Central nervous system and cardiac effects from long-acting amide local anesthetic toxicity in the intact animal model. Reg Anesth Pain Med. 2003 Jan-Feb;28(1):3-11. doi: 10.1053/rapm.2003.50014. PMID 12567336
- [Background] Mather LE, Copeland SE, Ladd LA. Acute toxicity of local anesthetics: underlying pharmacokinetic and pharmacodynamic concepts. Reg Anesth Pain Med. 2005 Nov-Dec;30(6):553-66. doi: 10.1016/j.rapm.2005.07.186. PMID 16326341
- [Background] Fredrickson MJ, Ball CM, Dalgleish AJ, Stewart AW, Short TG. A prospective randomized comparison of ultrasound and neurostimulation as needle end points for interscalene catheter placement. Anesth Analg. 2009 May;108(5):1695-700. doi: 10.1213/ane.0b013e31819c29b8. PMID 19372356
- [Background] Gautier P, Vandepitte C, Ramquet C, DeCoopman M, Xu D, Hadzic A. The minimum effective anesthetic volume of 0.75% ropivacaine in ultrasound-guided interscalene brachial plexus block. Anesth Analg. 2011 Oct;113(4):951-5. doi: 10.1213/ANE.0b013e31822b876f. Epub 2011 Aug 4. PMID 21821517
- [Background] Renes SH, van Geffen GJ, Rettig HC, Gielen MJ, Scheffer GJ. Minimum effective volume of local anesthetic for shoulder analgesia by ultrasound-guided block at root C7 with assessment of pulmonary function. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):529-34. doi: 10.1097/AAP.0b013e3181fa1190. PMID 20975468
- [Background] Marhofer P, Schrogendorfer K, Wallner T, Koinig H, Mayer N, Kapral S. Ultrasonographic guidance reduces the amount of local anesthetic for 3-in-1 blocks. Reg Anesth Pain Med. 1998 Nov-Dec;23(6):584-8. doi: 10.1016/s1098-7339(98)90086-4. PMID 9840855
- [Background] Ponrouch M, Bouic N, Bringuier S, Biboulet P, Choquet O, Kassim M, Bernard N, Capdevila X. Estimation and pharmacodynamic consequences of the minimum effective anesthetic volumes for median and ulnar nerve blocks: a randomized, double-blind, controlled comparison between ultrasound and nerve stimulation guidance. Anesth Analg. 2010 Oct;111(4):1059-64. doi: 10.1213/ANE.0b013e3181eb6372. Epub 2010 Aug 12. PMID 20705778
- [Background] Casati A, Baciarello M, Di Cianni S, Danelli G, De Marco G, Leone S, Rossi M, Fanelli G. Effects of ultrasound guidance on the minimum effective anaesthetic volume required to block the femoral nerve. Br J Anaesth. 2007 Jun;98(6):823-7. doi: 10.1093/bja/aem100. Epub 2007 May 3. PMID 17478453
- [Background] Riazi S, Carmichael N, Awad I, Holtby RM, McCartney CJ. Effect of local anaesthetic volume (20 vs 5 ml) on the efficacy and respiratory consequences of ultrasound-guided interscalene brachial plexus block. Br J Anaesth. 2008 Oct;101(4):549-56. doi: 10.1093/bja/aen229. Epub 2008 Aug 4. PMID 18682410
- [Background] Bernucci F, Gonzalez AP, Finlayson RJ, Tran DQ. A prospective, randomized comparison between perivascular and perineural ultrasound-guided axillary brachial plexus block. Reg Anesth Pain Med. 2012 Sep-Oct;37(5):473-7. doi: 10.1097/AAP.0b013e3182576b6f. PMID 22660484
- [Background] Imasogie N, Ganapathy S, Singh S, Armstrong K, Armstrong P. A prospective, randomized, double-blind comparison of ultrasound-guided axillary brachial plexus blocks using 2 versus 4 injections. Anesth Analg. 2010 Apr 1;110(4):1222-6. doi: 10.1213/ANE.0b013e3181cb6791. Epub 2010 Feb 8. PMID 20142336